CLINICAL TRIAL: NCT01163916
Title: A Multi-Center Post Marketing Observational Study to Characterize Demographics, Compliance, Tolerability and Safety in Patients With Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis Prescribed HUMIRA® (Adalimumab) as Part of Routine Clinical Care in Russia
Brief Title: Study to Characterize Demographics, Compliance, Tolerability and Safety in Patients With Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis Prescribed Adalimumab (Humira®) as Part of Routine Clinical Care
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Scientific Research Institute of Rheumatology, Moscow (Unknown); Almedis (Industry)
Responsible Party: Sponsor
Other Study IDs: P10-272
Record Dates: First submitted 2010-02-26; First posted 2010-07-16 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis
Keywords: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with RA, PsA and AS: Patients with Rheumatoid Arthritis (RA), Psoriatic Arthritis (PsA) and Ankylosing Spondylitis (AS) prescribed adalimumab as part of Routine Clinical Care in Russia.

SUMMARY:
The primary objective of this post-marketing observational study was to obtain data on the characteristics (patient age/gender; disease type, severity and duration; disease specific treatment history; current concomitant medications; other relevant medical history) of patients prescribed adalimumab (Humira®) for rheumatoid arthritis (RA), ankylosing spondylitis (AS) and psoriatic arthritis (PsA) as part of routine clinical care in Russia.

DETAILED DESCRIPTION:
This is a non-interventional, observational study in which adalimumab is prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication. No data currently exist that characterize patient types and adalimumab administration within the Russian population. Further, it is important to characterize the compliance, acceptability of patient self-injection, tolerability and safety profile of this therapy option with the routine clinical care.

The total follow-up for each participant was planned to be 12 months, with approximately 6 follow-up visits occurring at average intervals of 2-3 months. However, since this was an observational study, follow-up was performed according to routine clinical practice; for 127 participants the follow-up period consisted of more than 12 months and the maximum observation period lasted 18.2 months. Follow-up visits were designated sequential visit numbers (Visit 1-6), regardless of the time point at which they occurred.

ELIGIBILITY:
Inclusion Criteria:

Patients for whom adalimumab therapy is indicated according to product label and who meet the following criteria:

* Patients who are newly prescribed adalimumab therapy (no prior history of treatment with adalimumab) including patients with infliximab treatment history.
* Patients who completed Abbott sponsored interventional trials and are continuing treatment with commercial adalimumab thereafter.

Exclusion Criteria:

The following patients will not be included in the study:

* Patients who are being treated or will be treated with drugs at risk of interactions with adalimumab.
* Hypersensitivity to adalimumab
* Pregnancy
* Lactation
* Age below 18
* Infectious diseases including tuberculosis
* Patients currently participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis prescribed adalimumab as part of Routine Clinical Care in Russia.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey N Strugovschikov, MD, Study Director — Abbott Russia
Locations (43):
- Russia (43):
  - Site Ref # / Investigator 50728, Belgorod
  - Site Ref # / Investigator 50737, Chelyabinsk
  - Site Ref # / Investigator 50731, Izhevsk
  - Site Reference ID/Investigator# 29084, Kaliningrad
  - Site Reference ID/Investigator# 29163, Khanty-Mansiysk
  - Site Ref # / Investigator 50746, Khanty-Mansiysk
  - Site Ref # / Investigator 50736, Krasnogorsk
  - Site Ref # / Investigator 50727, Lipetsk
  - Site Ref # / Investigator 50723, Moscow
  - Site Ref # / Investigator 50725, Moscow
  - Site Ref # / Investigator 50742, Moscow
  - Site Ref # / Investigator 50743, Moscow
  - Site Ref # / Investigator 50724, Moscow
  - Site Ref # / Investigator 50739, Moscow
  - Site Ref # / Investigator 50732, Moscow
  - Site Ref # / Investigator 50738, Moscow
  - Site Ref # / Investigator 50744, Moscow
  - Site Reference ID/Investigator# 28989, Moscow
  - Site Reference ID/Investigator# 28990, Moscow
  - Site Reference ID/Investigator# 29195, Moscow
  - Site Reference ID/Investigator# 29482, Moscow
  - Site Reference ID/Investigator# 29483, Moscow
  - Site Ref # / Investigator 50740, Moscow
  - Site Ref # / Investigator 50733, Moscow
  - Site Ref # / Investigator 50745, Moscow
  - Site Ref # / Investigator 50741, Moscow
  - Site Reference ID/Investigator# 28956, Nizhnevartovsk
  - Site Reference ID/Investigator# 28968, Perm
  - Site Reference ID/Investigator# 28969, Perm
  - Site Reference ID/Investigator# 28957, Saint Petersburg
  - Site Reference ID/Investigator# 28997, Saint Petersburg
  - Site Reference ID/Investigator# 28999, Saint Petersburg
  - Site Reference ID/Investigator# 29001, Saint Petersburg
  - Site Reference ID/Investigator# 32403, Saint Petersburg
  - Site Ref # / Investigator 50729, Salekhard
  - Site Reference ID/Investigator# 29008, Surgut
  - Site Reference ID/Investigator# 32404, Tula
  - Site Reference ID/Investigator# 29095, Ulyanovsk
  - Site Ref # / Investigator 50734, V. Novgorod
  - Site Ref # / Investigator 50730, Vologda
  - Site Ref # / Investigator 50735, Voronezh
  - Site Ref # / Investigator 50726, Voronezh
  - Site Reference ID/Investigator# 6002, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis: Patients with rheumatoid arthritis prescribed adalimumab as part of routine clinical care in Russia.
- Psoriatic Arthritis: Patients with psoriatic arthritis prescribed adalimumab as part of routine clinical care in Russia.
- Ankylosing Spondylitis: Patients with ankylosing spondylitis prescribed adalimumab as part of routine clinical care in Russia.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Started | 126 | 35 | 91
Safety Population | 125 (One patient discontinued prior to receiving treatment with adalimumab due to absence of medication.) | 35 | 91
Completed | 96 (Completed 12-months treatment with adalimumab) | 31 (Completed 12-months treatment with adalimumab) | 71 (Completed 12-months treatment with adalimumab)
Not Completed | 30 | 4 | 20
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Other | 24 | 4 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis | Total
Number analyzed (Participants) | 126 | 35 | 91 | 252
Age Continuous [Mean (Standard Deviation); unit: years] | 47.0 (13.7) | 42.4 (12.6) | 36.2 (10.6) | 42.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 18 | 23 | 134
  Male | 33 | 17 | 68 | 118
Region of Enrollment [Number; unit: participants]
  Russian Federation | 126 | 35 | 91 | 252

OUTCOME MEASURES:

1. Primary Outcome: Characteristics of Patients Prescribed Adalimumab: Education Level
Description: Participants were asked to indicate their highest education level at the Baseline visit: secondary school, vocational school or college, university graduate, current university student, or other.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Rheumatoid Arthritis: Patients with rheumatoid arthritis, prescribed adalimumab as part of routine clinical care in Russia.
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 126 | 35 | 91
participants
  Secondary school | 21 | 2 | 5
  Vocational school/college | 34 | 9 | 26
  University degree | 64 | 19 | 51
  Current university student | 5 | 5 | 8
  Other | 2 | 0 | 1

2. Primary Outcome: Characteristics of Patients Prescribed Adalimumab: Occupation
Description: Participants were asked to indicate their occupation at the Baseline visit.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 126 | 35 | 91
participants
  Blue collar worker | 13 | 5 | 10
  Civil servant | 10 | 5 | 12
  White collar worker | 52 | 13 | 38
  Self-employed | 8 | 1 | 9
  Student | 7 | 4 | 4
  Retired | 21 | 4 | 4
  Other | 15 | 3 | 14

3. Primary Outcome: Characteristics of Patients Prescribed Adalimumab: Residence Status
Description: Participants were asked to indicate their residence status within the Russian Federation at the Baseline visit.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 126 | 35 | 91
participants
  Permanent | 113 | 33 | 88
  Temporary | 13 | 2 | 3

4. Secondary Outcome: Patient's Acceptability of Self-injections
Description: At each clinic visit participants were asked to rate the convenience of adalimumab injections. Possible options were "convenient," "inconvenient" and "unable to self-inject."
  The study follow-up period consisted of approximately 6 follow-up visits occurring at average intervals of 2-3 months, according to routine clinical practice.
  Acceptability data are reported by follow-up visit and by treatment regimen: 40 mg every other week or 40 mg once a week, as prescribed in accordance with local marketing authorization.
Time Frame: Data were collected at study follow-up visits (Visits 1-6) which occurred on average at 2-3 month intervals, up to a maximum of 18.2 months.
Population: The number of participants analyzed (251) represents the total number of participants in the safety set. The number of participants with available data at each follow-up visit were: Visit 1: 249; Visit 2: 246; Visit 3: 237; Visit 4: 205; Visit 5: 179; Visit 6: 135.
Measure: Number; unit: participants
Groups:
- Convenient: Participants who described the acceptability of adalimumab injections as "convenient."
- Not Convenient: Participants who described the acceptability of adalimumab injections as "not convenient."
- Need Assistance: Participants who were unable to self-inject.
- Missing: Participants for whom acceptability data were not available.
Arm/Group | Convenient | Not Convenient | Need Assistance | Missing
Number analyzed (Participants) | 251 | 251 | 251 | 251
participants
  Visit 1: 40 mg every other week | 168 | 10 | 71 | 0
  Visit 1: 40 mg once a week | 0 | 0 | 0 | 0
  Visit 2: 40 mg every other week | 172 | 7 | 63 | 0
  Visit 2: 40 mg once a week | 1 | 0 | 1 | 0
  Visit 2: Missing regimen data | 2 | 0 | 0 | 0
  Visit 3: 40 mg every other week | 177 | 7 | 49 | 0
  Visit 3: 40 mg once a week | 0 | 0 | 0 | 0
  Visit 3: Missing regimen data | 4 | 0 | 0 | 0
  Visit 4: 40 mg every other week | 155 | 3 | 45 | 0
  Visit 4: 40 mg once a week | 0 | 0 | 0 | 0
  Visit 4: Missing regimen data | 2 | 0 | 0 | 0
  Visit 5: 40 mg every other week | 137 | 1 | 39 | 0
  Visit 5: 40 mg once a week | 0 | 0 | 0 | 0
  Visit 5: Missing regimen data | 0 | 0 | 1 | 1
  Visit 6: 40 mg every other week | 105 | 1 | 27 | 0
  Visit 6: 40 mg once a week | 1 | 0 | 0 | 0
  Visit 6: Missing regimen data | 0 | 0 | 0 | 1

5. Secondary Outcome: Percentage of Participants With Missed or Delayed Injections
Description: Compliance with prescribed adalimumab therapy was assessed by the percentage of participants with missed injections and/or injections delayed by more than 7 days.
Time Frame: For the duration of the study (up to a maximum of 18.2 months).
Population: Safety set; the analysis only includes participants with non-missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 125 | 35 | 90
percentage of participants
  No missed or delayed injections | 55.2 | 57.1 | 56.7
  One missed or delayed injection | 21.6 | 11.4 | 21.1
  Two missed or delayed injections | 9.6 | 20.0 | 7.8
  Three or more missed or delayed injections | 13.6 | 11.4 | 14.4

6. Primary Outcome: Characteristics of Patients Prescribed Adalimumab: Marital Status
Description: Participants were asked to indicate their marital status at the Baseline visit.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 126 | 35 | 91
participants
  Married | 94 | 24 | 69
  Single | 32 | 11 | 21
  Missing | 0 | 0 | 1

7. Primary Outcome: Characteristics of Patients Prescribed Adalimumab: Disease Severity
Description: Disease severity was assessed by the physician as mild, moderate or severe, based on routine clinical practice.
Time Frame: Baseline
Population: Safety set.
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 125 | 35 | 91
participants
  Mild | 0 | 2 | 0
  Moderate | 44 | 14 | 31
  Severe | 81 | 19 | 60

8. Primary Outcome: Characteristics of Patients Prescribed Adalimumab: Duration of Disease
Description: Duration of disease was defined as the time from diagnosis until study entry.
Time Frame: Baseline
Population: Safety set
Measure: Median (Full Range); unit: months
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 125 | 35 | 91
months | 71.70 (81.91) [0.1 to 370.4] | 103.50 (110.02) [13.2 to 597.3] | 50.90 (79.47) [0.0 to 376.3]

9. Primary Outcome: Characteristics of Patients Prescribed Adalimumab: Other Disease Specific Treatment
Description: Data on other medications (methotrexate, non-steroidal anti-inflammatory drugs [NSAIDs], corticosteroids and other medications) taken for the participant's condition (rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis) were collected at the Baseline visit and at each follow-up visit throughout the study. Overall data are presented.
Time Frame: Baseline and at each follow-up visit (up to a maximum of 18.2 months).
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 125 | 35 | 91
participants
  Methotrexate | 96 | 23 | 20
  NSAIDs | 73 | 16 | 72
  Corticosteroids | 48 | 9 | 16
  Other medications | 82 | 18 | 65

10. Secondary Outcome: Duration of Treatment With Adalimumab
Description: Tolerability to adalimumab treatment was analyzed by the time on treatment until development of an adverse event leading to adalimumab discontinuation or until discontinuation from treatment for any other reason.
Time Frame: For the duration of the study (up to a maximum of 18.2 months).
Population: Safety set.
Measure: Median (Full Range); unit: weeks
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Number analyzed (Participants) | 125 | 35 | 91
weeks | 52.10 [0.1 to 74.0] | 52.90 [25.1 to 81.4] | 52.30 [10.3 to 78.0]

ADVERSE EVENTS:
Time Frame: Participants were followed for an average of 12 months with a maximum observation period of 18.2 months.
Arm/Group | Rheumatoid Arthritis | Psoriatic Arthritis | Ankylosing Spondylitis
Serious Adverse Events (participants affected / at risk) | 2/125 | 0/35 | 0/91
Other Adverse Events (participants affected / at risk) | 9/125 | 0/35 | 8/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis (N=125) | Psoriatic Arthritis (N=35) | Ankylosing Spondylitis (N=91)
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 1 | 0 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis (N=125) | Psoriatic Arthritis (N=35) | Ankylosing Spondylitis (N=91)
Respiratory tract infection viral (Infections and infestations) | 9 | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.